CLINICAL TRIAL: NCT07385235
Title: A Randomized, Open-label, Single-dose, Two-sequence, and Two-period Crossover Study to Evaluate the Pharmacokinetics and Safety Between the Administration of AD-115A and the Administration of AD-1151 for Healthy Subjects in Fasting State
Brief Title: Compare and Evaluate the Safety and PK Data of a Single Dose Administration of 'AD-115A' or 'AD-1151'
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-115BE-02
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Gastric Ulcer
MeSH Terms: conditions — Stomach Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1 : Reference Drug(Rebanex Tab), Period 2 : Test Drug(Revaprazan sulfate)
  Single-dose oral administration of AD-115A (200 mg tablet) in Period 1, followed by single-dose oral administration of AD-1151 (200 mg tablet) in Period 2.
  Interventions: Drug: AD-115A, AD-1151
- Sequence B (Experimental): Period 1 : Test Drug(Revaprazan sulfate), Period 2 : Reference Drug(Rebanex Tab)
  Single-dose oral administration of AD-115A (200 mg tablet) in Period 1, followed by single-dose oral administration of AD-1151 (200 mg tablet) in Period 2.
  Interventions: Drug: AD-115A, AD-1151

INTERVENTIONS:
Drug: AD-115A, AD-1151 — Single-dose oral administration of AD-115A or AD-1151 (200 mg tablet), according to randomized sequence.

SUMMARY:
The study compare and evaluate the safety and pharmacokinetic characteristics of a single dose administration of 'AD-115A' or 'AD-1151' in healthy adults.

DETAILED DESCRIPTION:
A randomized, open-label, single-dose, two-sequence, and two-period crossover study to evaluate the pharmacokinetics and safety between the administration of AD-115A and the administration of AD-1151 for healthy subjects in fasting state

ELIGIBILITY:
Inclusion Criteria:

* The Age equal to or greater than 19 in healthy volunteers at the time of screening visit
* Body mass index (BMI) between 18.0 kg/m2 and 30.0 kg/m2 at the time of screening visit

Exclusion Criteria:

* Individuals who have taken drugs that induce (e.g., barbiturates) or inhibit drug-metabolizing enzymes within 30 days prior to the start of the study (first dosing day), or have taken drugs that may affect this study within 10 days prior to the start of the study (first dosing day)
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2026-03-07 (Estimated); Study Completion 2026-03-16 (Estimated)

PRIMARY OUTCOMES:
Maximum concentration of drug in plasma (Cmax) | pre-dose to 24 hours
  Cmax of AD-115A
Area under the plasma concentration-time curve during dosing interval (AUCt) | pre-dose to 24 hours
  AUCt of AD-115A

CONTACTS AND LOCATIONS:
Locations (1):
- H PLUS YANGJI HOSPITAL, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No